CLINICAL TRIAL: NCT05721118
Title: Diagnostic Performances of Mandibular CBCT Versus DXA Gold-Standard in Bone Mineral Density Assessment and Osteoporosis Diagnosis.
Brief Title: Diagnostic Performances of Mandibular CBCT in Osteoporosis
Acronym: TOMOSTEOp
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TOMOSTEOp_AL_190123
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBCT and DXA exams performed in current practice in Nantes University Hospital — 40 patients will be enrolled in order to study DXA/CBCT acquisitions of 16 osteoporotic women vs 34 osteopenic/healthy women (Estimated osteoporotic rate = 20%)

SUMMARY:
In the last decade, there has been a shift towards Cone-Beam Computed Tomography (CBCT - regarding its low-dose radiation profile) in Dentistry/Implantology fields because it presents a more conclusive insight in the bone micro-architecture and cortical/trabecular bone structures assessment due to 3D acquisition higher resolution. Despite convergent and interesting preliminary results, most CBCT studies failed in highlighting a potential new osteoporosis diagnostic tool. TOMOSTEOp study aims to explore inter-relation between CBCT parameters and DXA Gold-Standard parameters in order to build resolutive explicative model of bone mineral density and test CBCT diagnostic performances.

DETAILED DESCRIPTION:
In the last decade, there has been a shift towards Cone-Beam Computed Tomography (CBCT - regarding its low-dose radiation profile) in Dentistry/Implantology fields because it presents a more conclusive insight in the bone micro-architecture and cortical/trabecular bone structures assessment due to 3D acquisition higher resolution. Despite convergent and interesting preliminary results, most CBCT studies failed in highlighting a potential new osteoporosis diagnostic tool. TOMOSTEO aims to explore inter-relation between CBCT parameters and DXA Gold-Standard parameters in order to build resolutive explicative model of bone mineral density and test CBCT diagnostic performances.

TOMOSTEOp study will analyze CBCT and DXA acquisitions of >65 years old post-menopausal women who performed contemporaneously (ie. maximum 3months delay) these 2 exams. Radiomorphometric (I/S/CTMI/CTI(S)/CTI(I)), Gray Values (cortical and trabecular) and Fractal Dimension Indexes will be measured on the whole mandibular arch, as well as cortical/trabecular thicknesses. Correlations and odds-ratio will be calculated regarding DXA parameters and T-scores (-2,5DS). Differences between osteopenic, osteoporotic and healthy women will be explored.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old post-menauposal women
* Contemporanean (ie. 3months) CBCT and DXA exams performed in Nantes University Hospital.

Exclusion Criteria:

* < 65 years old post-menauposal women
* CBCT and DXA exams interval superior to 3months.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Post-menauposal women
Study Population: >65 years old post-menopausal women who performed contemporaneously (ie. maximum 3months delay)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-08 (Estimated); Primary Completion 2023-03-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of diagnostic performances of CBCT multivariate explicative model of osteoporosis regarding DXA T-Score Gold-Standard (-2,5DS). | Day1 of retrospective CBCT/DXA acquisition analysis
  Sensitivity (Se), Specificity (Sp), Negative Predictive Value (NPV), Positive Predictive Value (PPV), AUC.

IPD SHARING:
Plan to Share IPD: No
Anonymized data. No sharing.

REFERENCES:
- [Derived] Legrand A, Autrusseau F, Bandiaky ON, Idiri K, Le Goff B, Amador G, Volteau C, Maugars Y, Soueidan A. Promising diagnostic performance of CBCT-based TOMOSTEOp algorithm in osteoporosis: toward a complementary populational screening tool managed by dentists? Osteoporos Int. 2023 Jun;34(6):1137-1138. doi: 10.1007/s00198-023-06724-8. Epub 2023 Mar 31. No abstract available. PMID 37000207